CLINICAL TRIAL: NCT01094353
Title: Randomised Trial of Ophira™ Minisling System and Unitape™ for the Treatment of Stress Urinary Incontinence in Women
Brief Title: A Comparative Study Minisling Versus Transobturator (TOT)Sling
Acronym: sui
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Livia Garcia Pascom, M.D., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ophira
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Female Stress Urinary Incontinence
Keywords: Urodynamic Stress urinary incontinence; Minisling; Ophira™; Unitape™
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Intervention Model Description: Clinical, prospective, single-center, randomized controlled trial comparing the efficacy and safety of a single-incision mini-sling and a transobturator midurethral sling for female stress urinary incontinence (SUI) treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants were randomly allocated to a single-incision mini-sling or a transobturator midurethral tape by a simple randomization procedure using a random number generator computer program. Randomization was performed at the moment of inclusion by a nurse blinded to women's histories. Group assign- ment was concealed in consecutively numbered, sealed, opaque envelopes that were opened in the operating room just before the procedure.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mini-sling (Active Comparator): The minisling Ophira™ is a new intervention therapeutic option for surgical treatment in women with stress urinary incontinence. It is made of polypropylene monofilament mesh, held between two self-anchoring polypropylene columns in a fishbone design connected to two delivering needles.
  Interventions: Procedure: Mini-sling
- Transobturator (Active Comparator): Transobturator sling Unitape™ is an outside-in approach therapeutic option for surgical treatment in women with stress urinary incontinence
  Interventions: Procedure: Transobturator

INTERVENTIONS:
Procedure: Mini-sling — The minisling is a new intervention therapeutic option for surgical treatment in women with stress urinary incontinence. It is made of polypropylene monofilament mesh, held between two self-anchoring polypropylene columns in a fishbone design connected to two delivering needles.
  Other Names: Mini-sling Ophira™
  Arms: Mini-sling
Procedure: Transobturator — Transobturator sling Unitape™ is an outside-in approach therapeutic option for surgical treatment in women with stress urinary incontinence
  Other Names: Transobturator Sling Unitape™
  Arms: Transobturator

SUMMARY:
A study to compare efficacy in surgical treatment for SUI (Stress Urinary Incontinence), tot with minisling.

DETAILED DESCRIPTION:
eligibility criteria was : female stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* clinical and urodynamic diagnosis of SUI in patients between 18 and 90 years

Exclusion Criteria:

* postvoid residual urine volume more than 100 ml, coagulation disorders, current urinary tract infection, sequelae of previous radiation therapy of the pelvis, anticoagulant therapy, vulvovaginitis, and anesthesia contraindication

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
to assess efficacy between tot with minisling in cure in women with stress urinary incontinence | one year
  to assess efficacy and safety of minisling and transobturator sling in treatment of female stress urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Ana LG Pascom, Pg, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] De Ridder D, Berkers J, Deprest J, Verguts J, Ost D, Hamid D, Van der Aa F. Single incision mini-sling versus a transobutaror sling: a comparative study on MiniArc and Monarc slings. Int Urogynecol J. 2010 Jul;21(7):773-8. doi: 10.1007/s00192-010-1127-z. Epub 2010 Mar 4. PMID 20204323
- [Derived] Djehdian LM, Araujo MP, Takano CC, Del-Roy CA, Sartori MGF, Girao MJBC, Castro RA. Transobturator sling compared with single-incision mini-sling for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2014 Mar;123(3):553-561. doi: 10.1097/AOG.0000000000000148. PMID 24499750